CLINICAL TRIAL: NCT02896439
Title: Protocol for Evaluation Effectiveness Monitoring Neurophysiological Per-operative in Surgery Traumatic Acetabular
Acronym: PESCIATIQUE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The principal investigator decided to stop the research.
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PESCIATIQUE
Record Dates: First submitted 2016-08-25; First posted 2016-09-12 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Surgery
Keywords: Traumatic; Acetabular
MeSH Terms: interventions — Neurophysiological Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurophysiological monitoring (Experimental)
  Interventions: Device: Neurophysiological MONITORING

INTERVENTIONS:
Device: Neurophysiological MONITORING — The neurophysiology team perform:
  * Implementation of the stimulation electrodes and collection (needle electrodes) SEP and EMG as described above.
  * Acquisition of data by the machine and the software Protektor® (Natus) in the following format:
  A PES stimulation every 10 minutes consistently. Meanwhile, important surgical time and known to be at risk for neurological injury will be noted and their exact schedule specified:
  * Establishment of a spacer or forceps in the greater or lesser sciatic notch
  * Traction layout
  For the ways of Kocher-Langenbeck, a collection of potential nerve sciatic trunk upstream of the critical region:
  * At the end of the incision
  * On the establishment of a spacer or forceps in the greater or lesser sciatic notch
  * When towing layout
  * At the end of the intervention

SUMMARY:
Pelvic fractures in which integrate the acetabulum fractures represent a risk of traumatic injury to the sciatic nerve trunk by stretching or section (1): Judet and Letournel reported a complication rate of around 6% (1). Fractures of the acetabulum strictly speaking are also providers of neurological complications with rates, significant, have recently been precisely detailed by a cohort study published by Lehmann et al. (2): In a series of 2073 patients, the authors reported an overall complication rate of neurological related to the initial trauma of the order of 4%. In this series, 1395 patients were operated with a rate of iatrogenic neurological complications of 2 to 3%. Regarding the first routes (and therefore the types of fractures), the Kocher-Langenbeck path is the path that leads to the greatest number of neurological complications: 3 to 4% in this series (2). However, this cohort study does not specify what truncal achievement it is. Obviously violations posterior acetabular are preferentially providers of sciatic injury while violations prior acetabular are more providers of obturator or femoral lesions. But this is not always the case. Moreover, this study does not specify the type or severity of neurological involvement.

DETAILED DESCRIPTION:
Methodology Design: This is an interventional study in routine care, prospective, single-center.

Main objective / secondary:

Primary objective :

To evaluate the sensitivity of the neurophysiological monitoring combining two specific new procedures to detect intraoperative complications on the sciatic trunk (by measuring potential with somatosensory storied collection of P15 and electromyographic recording with the potential of sciatic nerve in the popliteal fossa).

secondary objectives

Frequency of neurophysiological changes on the interventions of the acetabulum.

An anomaly being retained as:

* Interval prolongation N8-P15> 10%
* And / or decrease in the amplitude ratio P15 / N22> 50%
* And / or elongation of the latency of nerve potential> 10% of the value-operative Opré
* And / or reducing the amplitude of the nerve potential> 50% Correlation between the impact of changes neurophysiological intraoperative and
* The occurrence of postoperative neurological deficit:

  * motor deficit
  * and / or sensory deficit
  * territory of the sciatic trunk

Correlation between the incidence of intraoperative neurophysiological modifications and:

* The type of surgery
* The type of fracture

ELIGIBILITY:
Inclusion Criteria:

* Patients sent to the Hospital Group Service Paris Saint Joseph for surgical treatment of fractures of the acetabulum.
* Anterior and posterior surgical first Routes
* Major Patient
* Age <60 years

Exclusion Criteria:

* Known diabetes treated
* Previous history of spine surgery
* Sick antecedent the peripheral or central nervous system known

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2015-05-15 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2019-03-07 (Actual)

PRIMARY OUTCOMES:
Assessment of the score of electrophysiological intraoperative event | Day -1 before surgery
  The Score will be assessed between 1 to 3 (1= negative. 2= average, 3= good):
  * Potential to be studied subsequent stages, after averaging 500 successive traces to the following story:
    o popliteal Hollow: bipolar collection
  * Cathode medial, (1, 2 or 3 Point)
  * Anode side (1, 2 or 3 Point)
  * Recording the distal truncal response N8. (1, 2 or 3 Point)
  * Recorded values:
    * Latency N8 (1, 2 or 3 Point)
    * Amplitude o Basin bipolar collection,
  * Cathode: iliac crest to the stimulated nerve (1, 2 or 3 Point)
  * Anode: ipsilateral gluteal fold ((1, 2 or 3 Point)
  * Recording the P15 response. (1, 2 or 3 Point)
  * Recorded values:
    * Latency P15 (1, 2 or 3 Point)
    * P15 Amplitude (1, 2 or 3 Point)
    * Interval-P15 N8 (1, 2 or 3 Point) o Spinal cord dorsal low Bipolar collection
  * Cathode level D12 (1, 2 or 3 Point)
  * Umbilicus anode (1, 2 or 3 Point)
  * Saving the N22 potential. (1, 2 or 3 Point)

SECONDARY OUTCOMES:
Assessment of change of sensitivity: according to the quotation of the ASIA score | Day 2, Month 3, Month 6 et Month 12
Assessment of change of Pain (VAS) Visual Assessment Scale | Day 2, Month 3, Month 6 et Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume P RIOUALLLON, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided